CLINICAL TRIAL: NCT03549143
Title: Multicenter Observational Prospective Study to Describe Irritable Bowel Syndrome in the Russian Federation
Acronym: ROMERUS
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: EPIDI060
Record Dates: First submitted 2017-12-18; First posted 2018-06-07 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Irritable Bowel Syndrome; spasmolytics; mebeverine; Duspatalin
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IBS — No intervention, description of routine practice only

SUMMARY:
Observational Prospective Study to Describe Irritable Bowel Syndrome in the Russian Federation

DETAILED DESCRIPTION:
Awareness about the disease in Russia is extremely low both among doctors and especially among patients. To date there are no data on the prevalence of the disease in Russia. This is the first study to show patient profile, main trigger factors and concomitant diseases among patients with Irritable Bowel Syndrome (IBS) in Russia. Also treatment characteristics for these patients in Russia will be measured. This study fills a lack of scientific data about prevalence of IBS and additional information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-50 y.o
* Patients suffering from Irritable bowel syndrome (abdominal pain and changes in bowel habit) as defined by Rome IV criteria and the absence of any relevant structural disease
* Patient's written authorization to provide data for the program
* Patients who are able to input him/herself data into patients' part of Electronic Data Capture (EDC)

Exclusion Criteria:

Presence of alarm features:

* positive family history of colorectal cancer, inflammatory bowel disease, celiac disease
* rectal bleeding in the absence of documented bleeding hemorrhoids or anal fissures
* unintentional weight loss
* severe anemia (according to local laboratory reference values)
* Fever (> 37,5 degree Celsius)
* Night symptoms appearance

Other:

* Significant and progressive change in: enlargement of the liver, spleen, lymph nodes; ascites; palpable mass in the abdomen / pelvic
* Pregnancy or lactation or the inability to use adequate contraception during the study;
* Other conditions that made the patients participation impossible (by investigator judgment)
* Previous enrollment in any other clinical study during the course of this study, including participation in a study within 30 days prior to informed consent.
* Prescribed by Health Care Professional(s) (HCP) and being currently treated or having been treated with spasmolytics within the 3 months prior to entering the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult subjects, male and female, aged from 18 up to 50 years with symptoms potentially indicative of IBS according to ROME IV criteria
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-12-25 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with IBS according to Rome IV Diagnostic Criteria by sex | Baseline
Proportion of patients with IBS according to Rome IV Diagnostic Criteria by education | Baseline
Proportion of patients with IBS according to Rome IV Diagnostic Criteria by region of living | Baseline
Proportion of patients with IBS according to Rome IV Diagnostic Criteria by marriage status | Baseline
Proportion of patients with IBS according to Rome IV Diagnostic Criteria by type of IBS | Baseline

SECONDARY OUTCOMES:
Findings of routine examination | 6 months
  proportion of patients with confirmed IBS by routine examination among all patients met Rome IV criteria
Comorbidity | Baseline
  Proportion of patients with different diagnosis registered at baseline
Routine treatment regimens | Baseline, 6 months
  Proportion of patients received each treatment
Absolute score of the IBS symptoms measured by IBS-QoL scale | Baseline, 1, 2, 4, and 6 months
  Irritable Bowel Syndrome - Quality Of Life (IBS-QOL) questionnaire contains 34 questions assessed from 1 point = "not at all" till 5 point = "a great deal". The sum of all items is used to calculate the total score. All items are negative framed with the greatest response scale equaling the worst QoL. Scores for all items are transformed to a 0 to 100 scale, ranging from 0 (worst QoL) to 100 (best QoL).
Changes from baseline of the IBS symptoms measured by IBS-QoL scale | Baseline, 1, 2, 4, and 6 months
  Irritable Bowel Syndrome - Quality Of Life (IBS-QOL) questionnaire contains 34 questions assessed from 1 point = "not at all" till 5 point = "a great deal". The sum of all items is used to calculate the total score. All items are negative framed with the greatest response scale equaling the worst QoL. Scores for all items are transformed to a 0 to 100 scale, ranging from 0 (worst QoL) to 100 (best QoL). Positive change corresponds to better outcome.
Assesment by Global Patient Assessment scale | 1, 2, 4, and 6 months
  Global Patient Assessment contains one question to rate up patient's general complaints of GI-discomfort. A 5-point Likert scale is used as follow: 'symptom-free, markedly improved, slightly improved, unchanged, worse'.
Assesment by Physician Global Assessment scale | 1 and 6 months
  Physician Global Assessment contains one question to rate up patient's general complaints of GI-discomfort. A 5-point Likert scale is used as follow: 'symptom-free, markedly improved, slightly improved, unchanged, worse'.
Adherence to treatment | up to 6 months
  The national questionnaire of treatment compliance contains 5 questions with 4 answers each. The sum of all items is used to calculate the total score. The total score has the range from 0 (worst compliance) to 15 (best compliance).

CONTACTS AND LOCATIONS:
Locations (37):
- Russia (37):
  - City Clinical Hospital #8, Chelyabinsk
  - Railway Clinical Hospital, Irkutsk
  - City Clinical Hospital #4, Ivanovo
  - The First Republican Clinical Hospital of MoH UR, Izhevsk
  - Interregional Clinical Diagnostic Center, Kazan'
  - Medical Center "Dobryj Doctor", Kemerovo
  - Branch Hospital AT ST. Krasnodar JSC "RZD", Krasnodar
  - The Medical ON Group Lyubertsy, Lyubertsy
  - Institute of Health, Lyubertsy
  - SM-Clinic, Lyubertsy
  - Multidisciplinary Medical Clinic, Moscow
  - Research Institute of gastroenterology, Moscow
  - Medical Center 'Golden Orchid', Moscow
  - Outpatient Dpt of City Clinical Hospital #85, Moscow
  - Blokhin Oncology Center, Moscow
  - 9 MDC Ministry of Defense, Moscow
  - Medical Center on Timur Frunze Street, Moscow
  - MEDSI Clinic, Moscow
  - CP Litfonda, Moscow
  - Diamed Clinic, Moscow
  - MC Larmed, Moscow
  - Clinic 'Medic City', Moscow
  - MSMSU them. A. I. Evdokimov, Moscow
  - CPM LLC, Novosibirsk
  - LLC Multidisciplinary Medical Center ALTAME+, Odintsovo
  - LLC Industrial Medicine Clinic, polyclinic No1, Orenburg
  - Treatment and Rehabilitation Center No1, Rostov-on-Don
  - Medi Com LLC (SM-clinic), Saint Petersburg
  - LLC 'Avesta MDC-M', Saratov
  - Stavropol Regional Clinical Diagnostic Center, Stavropol
  - OKD Diagnostic Center, Surgut
  - Consulvative and Diagnostic Center Endos, Tyumen
  - Kuvatov RCH, Ufa
  - Diamed Llc, Vladivostok
  - MC Medic LLC, Yekaterinburg
  - MC Chance LLC, Yekaterinburg
  - LLC "Medical Center" Doctor Plus, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No